CLINICAL TRIAL: NCT02520089
Title: Comparison of Treatment of Humeral Shaft Pseudoarthrosis Between Bone Autograft Versus Platelet Rich Plasma. Randomized, Blinded Study
Brief Title: Humeral Shaft Pseudoarthrosis Treated With Bone Autograft Versus Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, MD, PhD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OR14-010
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Pseudoarthrosis
Keywords: platelet-rich plasma; bone grafting; pseudoarthrosis
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone autograft (Active Comparator): The investigator it will obtain bone autograft of iliac crest ipsilateral of each patient. And apply into the pseudoarthrosis focus at the moment of the fixation with a locking compression plates.
  Interventions: Procedure: bone autograft of iliac crest
- platelet rich plasma plus Bone autograft (Experimental): Other group of patients it will be extracted 40 mL of peripheric blood sample, and processed with a double-centrifugation technique to obtain 5 mL of platelet rich plasma, and collocated into the focus of pseudoarthrosis after standard fixation with locking compression plates and Bone Autograft of Iliac Crest.
  Interventions: Procedure: Platelet Rich Plasma plus bone autograft

INTERVENTIONS:
Procedure: bone autograft of iliac crest — The investigators will take bone autograft of iliac crest of the patient and then apply into the site of pseudoarthrosis, this graft have osteogenic, osteoinductive and osteoconductive properties
  Arms: Bone autograft
Procedure: Platelet Rich Plasma plus bone autograft — Sample of 40 mL of peripheric blood and processed to obtain 5 mL of platelet rich plasma, and collocated into pseudoarthrosis
  Other Names: Biomet GPS III; MTF Cascade
  Arms: platelet rich plasma plus Bone autograft

SUMMARY:
Patients with humeral shaft pseudoarthrosis is going to be treated with a standard protocol with a locking compression plate and bone autograft, and other group of patients treated with platelet rich plasma.

Posteriorly all the patients it will evaluated radiographically and with functional scales for a period of one year.

DETAILED DESCRIPTION:
Pseudarthrosis is a condition characterized by the absence of union from 3-4 months of the start of a fracture. It usually has symptoms manifested by pain and loss of function of the affected extremity. In addition to radiographic data with lack of consolidation in the fracture. The surgical indications in patients with pseudoarthrosis data are the presence of pain and the mobility of the fracture taking account the time evolution.

The humeral shaft fracture represent 3% of the general fractures, appearing around 66,000 cases per year in the United States. The conservative treatment with a brace has been used since the 1970's. Mostly of the humeral shaft fractures are managed with this option. Contraindications are those fractures which are bilateral or in polytraumatized patients who do not have the ability to roam.

Surgical treatment seeks to provide a stable fixation providing an early mobilization. The union of these fractures occurs in a period ranging from 12 to 24 weeks. The use of a Locking Compression Plate where there must be at least six cortical fixation on both fragments is actually recommended, besides is necessary applies also bone autograft to promote ossification has osteogenic, osteoinductive, and osteoconductive properties, with an radiographic union between the nineteen weeks.

The platelet-rich plasma (PRP) is obtained from a sample of autologous blood, and after processing it have growth factors that stimulate angiogenesis and cell proliferation. It has been used since 1990 to treat jaw fracture with bone autograft and tendon injury in rotator cuff with a good evolution. It has been bone consolidation from 8 to 24 weeks.

Preparation of platelet-rich plasma A 40-ml volume of whole blood was taken from the basilic or antecubital vein of the upper limb in sterile tubes and vacuum sealed with 3.8% sodium citrate as an anticoagulant. The samples were transported to the Tissue Engineering Laboratory of the Bone and Tissue Bank where they were centrifuged for 10 minutes at 1800 rpm to separate the cellular parts corresponding to the erythrocytes and leukocytes. The upper plasma layer was removed from each of the tubes (taking care not to remove the buffy coat) and collected into a 50-ml sterile conical polypropylene tube for a second centrifugation step for 12 min at 3400 rpm. The plasma supernatant, or platelet poor plasma, was removed, leaving a volume of 3 ml in which the platelets were resuspended. The 3 ml of PRP obtained was transferred to a sterile glass tube and vacuum sealed without anticoagulant. An aliquot of the final PRP was sent to the laboratory to quantify the number of platelets. Manipulation of the samples was performed in a sterile environment within a class II biosafety cabinet. Prior to the administration of PRP to the patient, activation of the platelets was induced by adding 0.45 ml of 10% calcium gluconate and inverting the sample several times to ensure a homogeneous mixture. Then, the activated PRP was aspirated with a 5-ml syringe for application to the patient using the technique described above after asepsis and the application of 2 ml of lidocaine into the application site.

The patient must sign the format of informed consent to the authorization of the surgery and the use of platelet-rich plasma.

After signing informed consent, will divide the patients in two randomized groups to make the comparative and longitudinal study. A control group of patients who will receive treatment with surgery on the basis of open reduction with locking compression plate and autologous bone of iliac crest. The experimental group of patients will receive the above-mentioned treatment more the application of plasma rich platelets at the level of the fracture focus.

After the surgery all the patients will be assessed at outpatient at 10 days for evaluation, pendulum exercises and the first radiographic evaluation. The patient will be attending consultation to continue his post-surgical evolution. During the follow-up visits, the radiographic extent of the bony callus was assessed via anteroposterior and lateral radiograph of the arm as follows grade 0, no identifiable bony callus; grade 1, primary bony callus formation with little or no new periosteal bone; grade 2, new periosteal bone formation on two sides of the humerus,; and grade 3, new periosteal bone formation on three or four sides of the humerus. The follow-up is for one year.

Sample size calculation Using a formula to test hypothesis and two mean difference, with a value of zα of 1.96 with significance level of 95 for two tails, and a value zβ of 0.84 with an output of 80, a sample was obtained of 7 participants per group, whereas an average of 19 weeks for group control with a standard deviation of 3 hoping to reduce up to 4 weeks the start of consolidation with the application of PRP.

ELIGIBILITY:
Inclusion Criteria:

* evolution of 3 months
* initial orthopedic management
* without mental illness

Exclusion Criteria:

* osteoporosis
* contralateral or ipsilateral fractures
* previous fracture in same place at least 3 month
* hematologic problems
* liver disease
* cardiac, renal or lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll EA, Schweppe M, Langfitt M, Miller AN, Halvorson JJ. Management of humeral shaft fractures. J Am Acad Orthop Surg. 2012 Jul;20(7):423-33. doi: 10.5435/JAAOS-20-07-423. PMID 22751161
- [Background] Lin J, Hou SM, Hang YS. Treatment of humeral shaft delayed unions and nonunions with humeral locked nails. J Trauma. 2000 Apr;48(4):695-703. doi: 10.1097/00005373-200004000-00018. PMID 10780604
- [Background] Pugh DM, McKee MD. Advances in the management of humeral nonunion. J Am Acad Orthop Surg. 2003 Jan-Feb;11(1):48-59. doi: 10.5435/00124635-200301000-00007. PMID 12699371
- [Background] Celebi L, Dogan O, Muratli HH, Yagmurlu MF, Yuksel HY, Bicimoglu A. [Treatment of humeral pseudarthroses by open reduction and internal fixation]. Acta Orthop Traumatol Turc. 2005;39(3):205-10. Turkish. PMID 16141726
- [Background] Khan SN, Cammisa FP Jr, Sandhu HS, Diwan AD, Girardi FP, Lane JM. The biology of bone grafting. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):77-86. PMID 15712985
- [Background] Ahmad Z, Howard D, Brooks RA, Wardale J, Henson FM, Getgood A, Rushton N. The role of platelet rich plasma in musculoskeletal science. JRSM Short Rep. 2012 Jun;3(6):40. doi: 10.1258/shorts.2011.011148. Epub 2012 Jun 19. PMID 22768374

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Autograft | Platelet Rich Plasma Plus Bone Autograft
Started | 12 | 11
Completed | 9 | 7
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Autograft | Platelet Rich Plasma Plus Bone Autograft | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (15.3) | 37.1 (10.2) | 38.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Stans Scale
Description: The evaluation of the radiographic extent of the bony callus (consolidation grade) will be assessed via anteroposterior and lateral radiograph of the arm and classified in different levels, as follows:
  * Grade 0, no identifiable bony callus .
  * Grade 1, primary bony callus formation with little or no new periosteal bone.
  * Grade 2, new periosteal bone formation on two sides of the humerus.
  * Grade 3, new periosteal bone formation on three or four sides of the humerus.
Time Frame: 9th month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone Autograft | Platelet Rich Plasma Plus Bone Autograft
Number analyzed (Participants) | 9 | 7
units on a scale | 2.7 (0.5) | 3.0 (0.0)

2. Secondary Outcome: Quick Disability of Arm, Shoulder and Hand
Description: It is designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. Where the better evaluation is equal to 0, and the worst evaluation is equal to 100.
Time Frame: 9th months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone Autograft | Platelet Rich Plasma Plus Bone Autograft
Number analyzed (Participants) | 9 | 7
units on a scale | 7.28 (11.3) | 5.32 (8.23)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bone Autograft | Platelet Rich Plasma Plus Bone Autograft
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes